CLINICAL TRIAL: NCT00816816
Title: Phase ⅡStudy of Neoadjuvant Chemotherapy Followed by Concurrent Chemoradiation for Stage ⅣAB Nasopharyngeal Carcinoma
Brief Title: Phase Ⅱ Study of Neoadjuvant Chemotherapy Followed by Concurrent Chemoradiation for Stage ⅣAB Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Department of Radiation Oncology,Cancer Hospital, Fudan University, Shanghai, China, Cancer Hospital, Fudan University, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-0703
Record Dates: First submitted 2009-01-02; First posted 2009-01-05 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2009-01

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Phase 2 Clinical Trial; NPC; neoadjuvant chemotherapy; concurrent chemoradiation
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Docetaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): All patients will receive docetaxel 75 mg/m2 on day 1; cisplatin 75 mg/m2 on day 1; and a continuous fluorouracil infusion at 500 mg/m2/d on days 1 through 5. Cycles are repeated every 21 days for a total of three cycles. Patients then will receive definitive radiotherapy with 3D-CRT or IMRT, and cisplatin (40mg/m2) weekly during external radiotherapy.
  Interventions: Drug: docetaxel, cisplatin, fluorouracil

INTERVENTIONS:
Drug: docetaxel, cisplatin, fluorouracil — neoadjuvant chemotherapy: docetaxel 75 mg/m2 on day 1; cisplatin 75 mg/m2 on day 1; and a continuous fluorouracil infusion at 500 mg/m2/d on days 1 through 5.
  concurrent chemotherapy:cisplatin 40 mg/m2 weekly.

SUMMARY:
The primary objective of this study is to determine the tolerance and overall survival in patients with stage ⅣAB NPC treated with neoadjuvant chemotherapy and concurrent chemoradiation.

Secondary objectives of the study are to evaluate the distant metastases free survival, and disease-free survival of patients with stage ⅣAB treated with this regimen

DETAILED DESCRIPTION:
Concurrent chemoradiation is the standard treatment for locally advanced NPC. The survival benefit gained from adding neoadjuvant chemotherapy to concurrent chemoradiation has never been defined. In the present trail, we hope to assess the tolerance and survival benefits of neoadjuvant chemotherapy followed by concurrent chemoradiation in patients with stage ⅣAB NPC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven differentiated non-keratinizing carcinoma, and undifferentiated carcinoma of the nasopharynx.
* Stage ⅣAB disease
* KPS >70
* Age between 18-70
* Patients should have adequate bone marrow function defined as an absolute peripheral granulocyte count (AGC) of > 2000 cells/mm3, platelet count of > 100,000 cells/mm3 (pre treatment without intervention). Bilirubin < 1.5 mg/dl, AST or ALT<2 x upper normal, serum creatinine<1.5mg/dl, creatinine clearance >50ml/min.
* No prior radiation treatment to the head and neck or any prior chemotherapy
* Patients with no prior malignancy (not include basal cell carcinoma of skin)

Exclusion Criteria:

* Evidence of metastases (below the clavicle or distant) by clinical or radiographic examinations.
* Prior radiotherapy to the head and neck region for any reason.
* Initial surgical treatment excluding diagnostic biopsy of the primary site or neck disease.
* Patients with previous or simultaneous primaries, excluding basal cell carcinoma or squamous cell carcinoma of skin.
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-12 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 and 5 years

SECONDARY OUTCOMES:
distant metastases free survival, and disease-free survival | 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lin Kong, MD, Principal Investigator — Department of Radiation Oncology, Cancer Hospital, Fudan University; Chaosu Hu, MD, Principal Investigator — Department of Radiation Oncology, Cancer Hospital, Fudan University
Locations (1):
- Department of Radiation Oncology, Cancer Hospital, Fudan University, Shanghai, China